CLINICAL TRIAL: NCT00941980
Title: Osteocel® Plus in Posterior Lumbar Interbody Fusion (PLIF): Evaluation of Radiographic and Patient Outcomes
Brief Title: Osteocel® Plus in Posterior Lumbar Interbody Fusion (PLIF)
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.OC-0809
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease
Keywords: biologics; fusion rates; PLIF; lumbar fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Osteocel Plus — biologic

SUMMARY:
This study is being conducted to determine the percentage of patients with solid spinal fusions after being treated with Osteocel Plus in a PLIF procedure. Due to the unique processing conditions, Osteocel Plus retains a high concentration of stem cells attached to the allograft bone matrix, so it is hypothesized that the fusion rate with Osteocel Plus will be comparable to published data for autograft. The Osteocel product family has already been used in approximately 20,000 cases worldwide.

DETAILED DESCRIPTION:
This is a prospective, non-randomized multi-center study to compare the use of Osteocel Plus in subjects who receive PLIF surgery at one or two levels. These subjects will present with degenerative conditions in the lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Subjects will receive Osteocel Plus during their PLIF operation. Subjects will be followed for 24-months following surgery to determine the number of study subjects that are solidly fused at or before 24 months postoperatively, and to determine the mean time to fusion. This data will be compared to published and/or retrospective data for autograft, synthetic ceramics and BMP.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent back and/or leg pain unresponsive to conservative treatment for at least six (6) months, unless clinically indicated earlier
2. Indicated for interbody fusion of one or two contiguous lumbar segments (L1 to S1)
3. Objective evidence of primary diagnosis must be confirmed by appropriate imaging studies
4. 18-70 years of age at the date of written informed consent
5. Able to undergo surgery based on physical exam, medical history and surgeon judgment
6. Expected to survive at least 2 years beyond surgery
7. Willing and able to return for post-treatment exams according to the follow-up called for in the protocol
8. Signed and dated Informed Consent Form

Exclusion Criteria:

1. Patient has a mental or physical condition that would limit the ability to comply with study requirements
2. Lumbar spine abnormality requiring treatment at more than two levels
3. Systemic or local infection; active or latent
4. Previous failed fusion at the operative level
5. Diseases that significantly inhibit bone healing (osteoporosis, metabolic bone disease, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease)
6. Undergoing chemotherapy or radiation treatment, or chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
7. Pregnant, or plans to become pregnant during the study
8. Subject is a prisoner
9. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contended)
10. A significant general illness (e.g., HIV, active metastatic cancer of any type) is present; subject is immunocompromised or is being treated with immunosuppressive agents
11. Participating in another clinical study that would confound study data

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the fusion rates of Osteocel Plus in one or two level(s) for PLIF subjects. | from pre-op to 24-month follow-up

SECONDARY OUTCOMES:
To evaluate the rate of complications for Osteocel Plus and compare to published and/or retrospective data for autograft or bone morphogenetic protein (BMP). | from pre-op to 24-month follow-up
To evaluate and compare radiographic outcome with respect to clinical outcome (function and pain). | from pre-op to 24-month follow-up
To evaluate and compare each outcome with respect to surgical time and blood loss. | from pre-op to 24-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Spine, Orthopaedic Rehabilitation Center, Lovelace Medical Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: NuVasive, Inc. — http://www.nuvasive.com